CLINICAL TRIAL: NCT03713138
Title: Therapeutic Role of Flax Seed for Poly Cystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allied Hospital Faisalabad (Other)
Responsible Party: Principal Investigator, Farhat Younas, Clinical Nutritionist, Allied Hospital Faisalabad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6099
Record Dates: First submitted 2018-10-13; First posted 2018-10-19 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Poly Cystic Ovary Syndrome
Keywords: Follicle stimulating hormone; Leutinizing hormone; Sex hormone binding globulin; Serum Prolactin; Flaxseed sachets; Lipid profile
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: Randomized controlled placebo trial
Who Masked: Participant
Masking Description: Single-blinded trial, Intervention and placebo given
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Flaxseed powder (Experimental): Three different quantities of flax seed powder were intervened to the subjects. One group was given 15 grams of flax seed a day. Second group was given 20 grams and third group was given 25 grams off lax seed a day.
  Intervention/ Dietary Supplement:
  Flax seed powder
  Three different quantities of flax seed powder were intervened to the subjects. One group was given 15 grams of flax seed a day. Second group was given 20 grams and third group was given 25 grams off lax seed a day.
  Other Name: intervention
  Interventions: Dietary Supplement: flaxseed powder
- Control group; Comparison group (No Intervention): The controlled group was given no intervention. No intervention was done to this group.
  Three different quantities of white flour were intervened to the subjects. One group was given 15 grams of white flour a day. Second group was given 20 grams and third group was given 25 grams of white flour a day.

INTERVENTIONS:
Dietary Supplement: flaxseed powder — Three different quantities of flax seed powder were intervened to the subjects. One group was given 15 grams of flax seed a day. Second group was given 20 grams and third group was given 25 grams off lax seed a day.
  Other Names: Intervention
  Arms: Intervention Flaxseed powder

SUMMARY:
The study was conducted to determine the therapeutic role of flax seed for Poly cystic ovary syndrome. A sample of 100 subjects were collected. The subjects were from various age group ranging from 18 to 45 years. Subjects showing the signs, symptoms, biochemical, and clinical parameters of the diseases were included in the study. Three different quantities of flax seed were introduced to the subjects for 90 days.

Objectives:

1. To assess the nutritional status of Poly cystic Ovary Syndrome patients
2. To determine the therapeutic role of flax seed for PCOS patients

Material and method: The level of follicle stimulating hormone, leutinizing hormone, sex hormone binding globulin, serum prolactin, ultrasound were analyzed. To determine the side effects of the flax seed, the liver-enzymatic, lipid profile, and renal tests were conducted.

DETAILED DESCRIPTION:
Material and methods

Study Population:

The data were collected from the Allied Hospital. All Females of ages 18 to 45 years, having PCOS attending the OPD of Allied Hospital was taken as the study population. Efficacy trials were conducted on the patients of PCOS, including females of age 18-45 years. They were divided into different groups (as per no. of selected treatments along with the control). Ten subjects left the study and were replaced. The project was approved by the ethical review committee.The feeding study was conducted with the cooperation of Allied Hospital. The study protocol was discussed with medical professionals and finalized after through technical suggestions.

Selection of subjects and Study Design

The patients were assorted randomly into four groups, 25 in each, namely control (T0),

A total 100 female subjects were included in the study as under A) Control: To: 25 B) Experimental groups (PCOS): 75

1. T1: 25
2. T2: 25
3. T3: 25

Inclusion Criteria:

All females of age 18 to 45 having PCOS

Women showing the presence of two out of three features (Oligo- or anovulation, hyper-androgenism, or poly cystic ovaries (Ovarian volume >10cc, 12 or more peripherally located follicles 2-9 mm in diameter or hypo-echoic enlarged ovaries with hyper-echoic central stroma in USG). Patients on Metformin (used for insulin resistance)

Exclusion Criteria:

* Females under 18 and above 45 years of age
* Those on any other medical therapy
* Pregnant and lactating women
* Those with a history of allergy to flax seed
* Women on anti-platelet and fibrinolytic drugs
* Women showing signs of PCOS but showing normal ovaries on ultrasound

Study Design

It was literature review based intervention study. The selected population for intervention purposes was studied twice, i.e. before and after the intervention of the selected nutraceutical. The same subjects were studied once again after one month of stopping the intake of selected nutraceutical. The change in results has confirmed the effects of the intervention.

This has been divided into four phases.

1. Phase-1:Assessment of the nutritional Status in PCOS
2. Phase -2:Development of nutraceutical (flaxseed sachets)
3. Phase -3:Intervention to study the effect of selected nutraceutical
4. Phase-4:Blood Analysis

   The procedure adopted in each of the above phases is explained as follows:

   Phase-1: Assessment of the nutritional status of selected patients

   This was done in Allied Hospital, patients attending OPD of gynecology ward was assessed for nutritional status. Following parameters were studied for this purpose
   * Family History
   * Medical history
   * Physical signs (thyroid gland, height, weight, skin, hair, breasts, belly, and BMI)
   * Menstrual cycle detail (menarche, frequency, duration, and severity)
   * History of dysmenorrhea
   * Ferriman-Gall way scoring for hirsutism
   * Marital status, parity, and difficulty in conception

   Phase -2: Development of Nutraceutical (flaxseed sachets)

   Procurement of raw materials Preparation of flax seed powder Preparation of flax seed sachets

   Phase-3: Intervention

   An acceptable number of human volunteers were selected keeping in view all ethical considerations. (25 in each group)
   1. Control group (To)
   2. Flaxseed (5 g) xTTS = 15 g/day (T1)
   3. Flaxseed (6.6 g) x TTS = 20 g/day (T2)
   4. Flaxseed (8.3 g) xTTS = 25 g/day (T3)

   The flaxseed powder from the selected treatments was given daily for a period of 12 weeks. The dietary history of the subjects was monitored with the help of a Food Diary on a weekly basis. Education/counselling were provided to the patients for necessary compliance with the restricted diet for PCOS.

   Phase-4: Blood Analysis and Ultrasound

   After three months of intervention blood tests: follicle stimulating hormone (FSH), Luteinizing hormone (LH) thyroid stimulating hormone (TSH), serum prolactin, and ultrasound will be repeated.

   Biochemical assays

   Follicles stimulating hormone

   The blood sample was taken to determine the quantitative level of serum follicles stimulating hormone (FSH) in patients fed with flaxseed powder by following the Immuno-enzymatic calorimetric method (ELISA).

   Luteinizing hormone

   The blood sample was taken to determine the quantitative level of serum luteinizing hormone (LH) in patients fed with flaxseed powder by following the Immuno-enzymatic calorimetric method.

   Sex hormone binding globulin

   The serum sex hormone binding globulin hormone (SHBG) in patients fed with flaxseed powder was determined by following the Rosner's method.

   Prolactin

   The serum sex prolactin level in patients fed with flaxseed powder was determined by following the radio-immunological method.

   Thyroid stimulating hormone

   The thyroid stimulating hormone (TSH) level in patients fed with flaxseed powder was performed to determine the thyroid gland functioning by following the third-generation non-isotopic method.

   Liver Function Test

   Alkaline Phosphatase (ALP)

   The activity of alanine phosphatase in the plasma was determined by using enzyme-linked immune-sorbent assay kit method.

   Aspartate Aminotransferase (AST)

   The activity alanine transferase in the plasma was determined by using di-nitrophenyl hydrazine (DNPH) method using Sigma kits 59-50 and 58-50 under the conditions.

   Alanine Aminotransferase (ALT)

   The activity alanine aminotransferase in the plasma was determined by using enzyme-linked immune-sorbent assay kit method.

   Lipid Profile

   Low-density lipoprotein (LDL)

   Serum low-density lipoprotein (LDL) was estimated by following the protocol of Vinson.

   High-density lipoprotein (HDL)

   The high-density lipoprotein (HDL) was assessed by HDL-Cholesterol precipitation.

   Triglyceride

   The triglyceride in the collected serum was determined by liquid triglyceride (GPO-PAP) method.

   Renal Function Tests

   Urea

   The flax seed fed patients were diagnosed with urea content by GLDH method with the help of commercial kit.

   Creatinine

   The blood creatinine of the patients fed on flax seed powder was determined by the Jaffe method using creatinine commercial kit.

   Follicles present in ovaries

   Ultrasound of the ovaries was carried out to check the number of follicles present in the ovaries.

   Size of the ovaries

   The size of the ovaries of patients fed with flax seed powder was also checked in ultrasound.

   Fasting blood glucose level

   The blood sample was taken to check the fasting blood glucose level. The sample was taken eight hours after eating. Fasting blood glucose level as determined by glucose dye oxido-reductase mediator reaction which is specific for glucose by glucometer Accuchek active.

   Research instruments
   1. Questionnaire: For screening/nutritional assessment of PCOS patients
   2. Hormonal analysis: Follicle stimulating hormone (FSH), luteinizing hormone (LH) thyroid stimulating hormone (TSH), Sex Hormone binding globulin (SHBG), and serum prolactin.
   3. Biochemical assay: ALP, ALT, AST, urea, Creatinine, Fasting blood glucose level, LDL, HDL, and triglyceride.

   Ethical Considerations:Written ethical approval was taken from the management of the concerned hospital and HOD of Gynecology department of the selected hospital. The consent was taken from the subjects after explaining the purpose of the study and after getting their consent for their menstrual cycle history, blood tests and ultrasound.

   Statistical analysis

   The data were subjected to statistical analysis by using the SPSS statistical package, analysis of variance (ANOVA) and least significant difference (LSD) was used to determine any significant difference among the treatments at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* • All females of age 18 to 45 having PCOS

  * Women showing the presence of two out of three features (Oligo- or anovulation, hyper-androgenism, or polycystic ovaries (Ovarian volume >10cc, 12 or more peripherally located follicles 2-9 mm in diameter or hypo-echoic enlarged ovaries with hyper-echoic central stroma in USG)
  * Patients on Metformin (used for insulin resistance)

Exclusion Criteria:

* • Females under 18 and above 45 years of age

  * Those on any other medical therapy
  * Pregnant and lactating women
  * Those with a history of allergy to flaxseed
  * Women on antiplatelet and fibrinolytic drugs
  * Women showing signs of PCOS but showing normal ovaries on ultrasound

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Follicle stimulating hormone (mIU/MI) | 3 months
  The blood sample was taken to determine the quantitative level of serum follicles stimulating hormone (FSH) in patients fed with flaxseed powder by following the Immuno-enzymatic calorimetric method (ELISA).
Leutinizing Hormone (mIU/MI) | 3 months
  The blood sample was taken to determine the quantitative level of serum luteinizing hormone (LH) in patients fed with flaxseed powder by following the Immuno-enzymatic calorimetric method (ELISA-ALPCO)
Sex hormone binding globulin (mg/dL) | 3 months
  The serum sex hormone binding globulin hormone (SHBG) in patients fed with flaxseed powder was determined by following the Rosner's method.
Serum Prolactin (ng/ml) | 3 months
  The serum sex prolactin level in patients fed with flaxseed powder was determined by following the radio-immunological method.

SECONDARY OUTCOMES:
blood sugar fasting (mg/dL) | 3 months
  The blood sample was taken to check the fasting blood glucose level. The sample was taken eight hours after eating. Fasting blood glucose level as determined by glucose dye oxido-reductase mediator reaction which is specific for glucose by glucometer Accuchek active
Thyroid stimulating hormone (Ml/L) | 3 months
  The thyroid stimulating hormone (TSH) level in patients fed with flaxseed powder was performed to determine the thyroid gland functioning by following the third-generation non-isotopic method.

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Mahmood, MPhill, Study Director — Akuwat
Locations (1):
- Allama Iqbal Open University, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No